CLINICAL TRIAL: NCT07132450
Title: Current Practice of Sedation and Analgesia Bundled Strategies Among ICU Nurses: A National Cross-sectional Survey
Brief Title: Sedation and Analgesia Bundled Strategies Among ICU Nurses
Status: Not yet recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ZWQ21886-2025-427
Record Dates: First submitted 2025-08-04; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2024-11

CONDITIONS: Sedation and Analgesia; Delirium; Family Invlovement/Empowerment; Early Mobilization
MeSH Terms: conditions — Agnosia; Delirium; Empowerment

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICU nurses: ICU nurses work form 28 provinces and cities in China. The inclusion criteria entailed: (1) possessing a valid nurse professional qualification certificate, and (2) having worked in an ICU for a minimum of one year. Conversely, the exclusion criteria stipulated: (1) nurses who were not working in the ICU during the study period, and (2) those in rotation or undergoing advanced training.

SUMMARY:
This is a prospective observational study to investigate the current clinical practice status of sedation and analgesia bundled strategies among ICU nurses

DETAILED DESCRIPTION:
Since the development of critical care medicine, analgesia and sedation management strategies have occupied an increasingly crucial position in the treatment of critically ill patients. Previous studies indicate that the traditional notion that deep sedation allows patients to "rest" and avoid painful memories is misguided. Deep sedation not only fails to deliver the anticipated benefits but is highly likely to prolong the patient's recovery cycle and impede physical recuperation.In actual intensive care practice, precisely and meticulously controlling the depth of analgesia and sedation is fundamental to ensuring patient comfort and the safety of clinical procedures. If the patient is in a state of pain and agitation, it is highly probable to trigger a series of severe adverse consequences, such as chronic pain and post-traumatic stress symptoms. These symptoms may persist long after the patient is discharged from the ICU, causing sustained damage to their physical and mental health. Simultaneously, the pain response significantly increases the patient's oxygen demand and the release of endogenous catecholamines, subsequently leading to a hypermetabolic state. These physiological changes will undoubtedly markedly delay the patient's recovery process.

Current critical care practices commonly emphasize the use of multimodal analgesia regimens, frequent assessment of patients' pain and sedation levels, and the implementation of light sedation using short-acting agents whenever feasible. These scientifically validated measures collectively form the influential ABCDEF bundled strategy (namely: Assessment, prevention, and management of pain; Both Spontaneous Awakening Trials (SATs) and Spontaneous Breathing Trials (SBTs); Choice of analgesia and sedation; Delirium assessment, prevention, and management; Early mobilization and Exercise; Family engagement and empowerment) .However, despite the significant theoretical advantages of the ABCDEF bundled strategy, its progress in actual clinical implementation has been slow. The sudden outbreak of the COVID-19 pandemic, in particular, delivered a substantial blow to healthcare systems. Compounded by multiple challenges such as drug shortages, resource constraints, and insufficient staffing, it has led to some irrational shifts in clinical practice. For instance, the proportion of deep sedation strategies has increased, the use frequency of benzodiazepines has risen, and compliance with daily sedation interruption has significantly decreased. These adverse changes severely compromise patient monitoring quality, subsequently exerting an extremely detrimental impact on patient prognosis.

Therefore, this study aims to gain insights into the current implementation status of the analgesia and sedation bundled strategy for critically ill patients among ICU nurses in China, as well as the underlying barriers. Its goal is to provide a robust and reliable scientific basis for optimizing the management strategies for critically ill patients and enhancing treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. possessing a valid nurse professional qualification certificate,
2. having worked in an ICU for a minimum of one year.

Exclusion Criteria:

1. nurses who were not working in the ICU during the study period
2. those in rotation or undergoing advanced training. All subjects must sign the online informed consent form before filling out the questionnaire.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU nurses work from 28 provinces and cities in China
Sampling Method: Non-Probability Sample
Enrollment: 228 (Estimated)
Dates: Start 2025-08-30 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Scale of management of pain | Day 1
  A self-designed scale is used to evaluate the nurses clinical practice of the assessment, prevention and management of pain.The counting data is represented by frequency and percentiles. Items include:Use any scale to assess the patient's pain，Scale Commonly used for pain assessment，Administer analgesia to the patient in advance before nursing operations (such as venipuncture, exercise, etc.)，Work in accordance with the standardized procedures for pain management in the ICU.
Scale of both spontaneous awakening tests(SATs) and spontaneous breathing tests(SBTs) | Day 1
  A self-designed scale is used to evaluate the nurses clinical practice of the SATs and SBTs experiment.The counting data is represented by frequency and percentiles. Project include:Frequency of the SATs conducted every day、Perform SBTs for mechanically ventilated patients every day、Work in accordance with the standardized procedures of "Awakening and Breathing" in the ICU、Role in SATs/SBTs.
Scale of choice of sedation and analgesia | Day 1
  A self-designed scale is used to evaluate the clinical practice of nurses choice of sedation and analgesia. The counting data is represented by frequency and percentiles.Projects include:Scales commonly used to evaluate the sedation status、Work in accordance with the standardized procedures for sedation management in the ICU、Maintain the minimum sedation limit for the patient or no sedation strategy、Advise intensivists to reduce the use of benzodiazepines.
Scale of delirium: assessment, prevention and management | Day 1
  A self-designed scale is used to evaluate the clinical practice of nurses in the assessment, prevention, and management of patients' delirium. The counting data is represented by frequency and percentiles.Projects include：Monitor delirium for ICU patients regularly、Scales commomly used to assess delirium、Role in delirium assessment、Pay attention to the underlying causes of delirium in patients、Examinations often being paid attention to understand the causes of delirium in patients、Measures are often taken to prevent delirium、Provide earplugs to patients for use、Non-pharmacological interventions to promote patient sleep、Advise intensivists to use drugs to promote sleep、Work in accordance with the standardized procedures for delirium management in the ICU、Provide cognitive stimulation to ICU patients
Scale of early mobility and exercise | Day 1
  A self-designed scale is used to evaluate the clinical practice of nurses in the e early mobility and exercise. The counting data is represented by frequency and percentiles.Projects include：Evaluate the patient's ICU-AW、Common assessment tools used for ICU-AW、Implement early activities for ICU patients、ICU activity scales used for goal-directed early activity (e.g., SOMS, PFIT, CPAx, FSS-ICU)、Types of exercises offered for ICU patients、AS a member of the ICU rehabilitation team.
Scale of family involvement and empowerment | Day 1
  A self-designed scale is used to evaluate the clinical practice of nurses in the patients' family involvement and empowerment. The counting data is represented by frequency and percentiles.Projects include：Explain delirium to family members、Enhance the delirium knowledge of family members through brochures or educational materials、Involve family members in delirium management、Strategies commonly used for family participation and empowerment.

SECONDARY OUTCOMES:
Scale of barriers in the current practice of bundled strategies in ICU nurses | Day 1
  A self-designed scale is used to exploring the barriers in the current practice of bundled strategies in ICU nurses.The counting data is represented by frequency and percentiles.Projects include：Barriers related to patients and family members、Barriers related to clinical medical staff、Barriers related to the bundled strategies、Barriers related to ICU environment.

IPD SHARING:
Plan to Share IPD: Undecided